CLINICAL TRIAL: NCT02863055
Title: Nintedanib as Maintenance Treatment of Pleural Malignant Mesothelioma (NEMO): a Randomized Double Blinded Phase II Study of the EORTC Lung Cancer Group
Brief Title: Nintedanib as Switch Maintenance Treatment of Pleural Malignant Mesothelioma
Acronym: NEMO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of scientific relevance (change in the treatment landscape) and poor recruitment
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EORTC-08112
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: MPM; Unresectable; Phase II; Randomized; Maintenance
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nintedanib (Experimental): 200 mg twice a day per os
  Interventions: Drug: Nintedanib
- Placebo (Placebo Comparator): Placebo match twice a day per os
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nintedanib — Nintedanib 200 mg administered twice daily
  Arms: Nintedanib
Drug: Placebo — Matching placebo administered twice daily
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, 1:1, double blinded phase II trial. Patients with unresectable malignant pleural mesothelioma (MPM) will be randomized between arm A: nintedanib and arm B:placebo

DETAILED DESCRIPTION:
This is a multicenter, prospective, double blinded, randomized, two-arm phase II trial aiming to evaluate nintedanib treatment as switch maintenance in patients with unresectable MPM.

After signing of the informed consent and upon confirmation of all eligibility criteria, patients will be randomized 1:1 to:

* Arm A: twice daily nintedanib at a dose of 200 mg until progression or unacceptable toxicities.
* Arm B: matched placebo.

Response evaluation will be performed through CT scans every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of unresectable Malignant Pleural Mesothelioma (MPM);
* Response or Stable disease according to modified RECIST criteria [48] after first line platinum-pemetrexed chemotherapy for 4-6 cycles;
* Last platinum chemotherapy dose administered within 60 days (i.e. randomization must occur within 60 days from the last dose of the last cycle of platinum-pemetrexed chemotherapy);
* Age >18 years;
* ECOG performance status (PS) 0-2;
* Life expectancy of at least 12 weeks in the opinion of the investigator;
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to start of first dose

Exclusion Criteria:

* prior systemic anticancer therapy including cytotoxic therapy or immune-checkpoint inhibitor, for MPM, other than first line platinum-based doublet chemotherapy;
* previous extra-pleural pneumonectomy (other forms of previous surgery eg pleurectomy are acceptable);
* previous Vascular Endothelial Growth Factor (VEGF) inhibitors (eg bevacizumab, sorafenib, etc);
* treatment with other investigational drugs or treatment in another clinical interventional trial within the past 4 weeks before start of therapy or concomitantly with the trial;
* patients that, in the opinion of the investigator, have reduced performance status by 2 ECOG levels (e.g. PS 0 to 2 or PS 1 to 3) from beginning to completion of 1st line chemotherapy;
* radiotherapy (with the exception of palliative radiotherapy) during study or within 4 weeks of start of study drug;
* known brain metastasis or lepto-meningeal disease. Patients with suspicious neurological symptoms should undergo a CT scan/MRI of the brain to exclude brain metastasisNo active brain metastases (e.g. stable for < 4 weeks;, no adequate previous treatment with radiotherapy;, symptomatic, requiring treatment with anti-convulsants; dexamethasone therapy will be allowed if administered as stable dose for at least one month before randomization); patients with suspicious neurological symptoms should undergo a CT scan/MRI of the brain to assess brain metastasis;
* leptomeningeal metastases;
* significant weight loss (> 10 %) within the past 6 weeks prior to treatment in the present trial;
* pre-existing clinically significant ascites and/or clinically significant pleural effusion;
* active or history of bleeding complications that would prevent anti-angiogenic therapy
* centrally located tumors with radiographic evidence (CT or MRI) of local invasion of major blood vessels; typical mediastinal pleural involvement with mesothelioma remains eligible;
* clinically active cancer other than mesothelioma within 5 years prior to start of study treatment;
* radiographic evidence of cavitatory or necrotic tumors;
* unstoppable use of therapeutic anticoagulation (except low dose heparin and/or heparin flush as needed for maintenance of an indwelling intravenous device) or antiplatelet therapy (except for chronic low-dose therapy with acetylsalicylic acid =325mg per day);
* clinically significant cardiovascular diseases (i.e. hypertension not controlled by medical therapy, unstable angina, history of myocardial infarction within the past 6 months, congestive New York Heart Association (NYHA) II, serious cardiac arrhythmia, clinically significant pericardial effusion)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-02-04 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 6 months
  From randomization until progression or death

SECONDARY OUTCOMES:
Overall survival | 12 months
  From randomization until progression or death
Overall Response Rate | 6 months
  Response according to modified RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Popat, PhD, MD, Principal Investigator — Royal Marsden NHS Foundation Trust; Omar Abdel-Rahman, MD, Principal Investigator — Ain Shams University
Locations (9):
- Belgium (2):
  - UZ Antwerpen, Antwerp
  - UZ Gent, Ghent
- Ospedale San Paolo, Milan, Italy
- United Kingdom (6):
  - Manchester University NHS Foundation Trust - UHSM-Wythenshawe Hospital, Wythenshawe, Manchester
  - Royal Marsden Hospital, Chelsea
  - Royal Marsden Hospital - Kingston, Kingston
  - Sheffield Teaching Hospitals NHS Foundation Trust - Weston Park Hospital, Sheffield
  - NHS South Tyneside-South Tyneside District Hospital, South Shields
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No